CLINICAL TRIAL: NCT04969302
Title: Examination of the Effect of Skin Antisepsis With Pre-heated Povidone Iodine on Surgical Site Infections: A Quasi-Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Kerem Yıldız, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 19/21
Record Dates: First submitted 2021-06-26; First posted 2021-07-20 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Surgical Site Infections
Keywords: Povidone Iodine; Skin antisepsis; Abdominal Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Skin preparations will performe using Povidone 10% 1000 mL solution (Turkuaz Chemistry, İstanbul, Turkey) Povidone-iodine will heat to 37°C using a gel warmer (KGW-1 Keewell Medical Technology, Foshen, China) in the warm group.
  The day before the operation, the patient will be met and informed about the study and verbal and written consent will be obtained stating that they are willing to participate in the study.
  The weight tracking of the patients will be determined using a digital weight meter provided by the researcher. Patient evaluation will be made with NRS-2002 in terms of malnutrition risk.
  Antibiotic prophylaxis of 1000 mg available in the operating room will be administered 30-60 minutes before the operation.
  Before the incision, a wound culture sample will be taken with sterile transport swap and sent to the laboratory for culture study.
  Interventions: Diagnostic Test: Follow-up
- Control Group (No Intervention): Skin preparations will performe using Povidone 10% 1000 mL solution (Turkuaz Chemistry, İstanbul, Turkey) Povidone-iodine will heat to 20°C using a gel warmer (KGW-1 Keewell Medical Technology, Foshen, China) in the room heat group.
  The day before the operation, the patient will be met and informed about the study and verbal and written consent will be obtained stating that they are willing to participate in the study.
  The weight tracking of the patients will be determined using a digital weight meter provided by the researcher. Patient evaluation will be made with NRS-2002 in terms of malnutrition risk.
  Antibiotic prophylaxis of 1000 mg available in the operating room will be administered 30-60 minutes before the operation.
  Before the incision, a wound culture sample will be taken with sterile transport swap and sent to the laboratory for culture study.

INTERVENTIONS:
Diagnostic Test: Follow-up — The primary outcome of this study was SSI within 30 days of surgery, as defined by the Centers for Disease Control and Prevention. Secondary outcomes were identification of the causative organism, and investigation of clinical factors such as body mass index (BMI), operation time, days of hospitalization, etc. that may be associated with SSI.
  All patients were followed up for SSI until discharge from hospital and at the outpatient visits. SSI surveillance data forms were used for the collection of primary and secondary outcome data.
  SSI rates and distribution of identified micro-organisms for each group will measured
  Arms: Intervention Group

SUMMARY:
Surgical Site Infections (SSI) develop as a complication of surgical care 30-90 days after surgery without implants and within 1 year after implanted operations. Despite advances in asepsis practices, sterilization methods, surgical technique and antibiotic prophylaxis, SSI is the most important cause of hospital stay, morbidity and even mortality. SSI, which constitutes approximately 20% of healthcare associated infections (HAI) all over the world, is also the HAI with the highest cost. Although it has been reported that 60% of the SSI can be prevented by using evidence-based guidelines, 2-5% of the operated patients develop SSI, the hospital stay of patients with SSI is 7-11 days longer, the risk of death increases 2-11 times, It was reported that the cause of death was direct SSI. In the United States of America (USA), SSI constitutes 31% of HAI, it is seen in 2-5% of inpatients, approximately 160,000-300,000 SSIs occur each year, the most common and costly HAI.Abdominal surgery; It includes the treatment of diseases of organs such as stomach, gall bladder, pancreas, spleen, liver, small intestine and large intestine. It has been reported that the incidence of SSIs after abdominal surgery is 15-25% higher than other types of surgery. In a study conducted by Alcan et al. (2020), 69.8% of nurses stated that they used Povidone Iodine as skin antisepsis. Wistrand et al. (2015) compared preoperative 36 ° C and room temperature 20 ° C Chlorhexidine Gluconate solutions, but reported that there was no difference in bacterial colonization and SSI rates. In their study in Turkey, Gezer et al. (2020) reported that the prevalence of SSI was significantly lower in the Povidone Iodine group heated to 37 ° C before surgery compared to the Povidone Iodine group applied at 25 ° C room temperature.

DETAILED DESCRIPTION:
This study was planned in accordance with a single blind randomized controlled full experimental study design to determine the effect of skin antisepsis with Povidone Iodine, which was heated at 37°C and at a room temperature of 20°C in the preoperative period, in reducing surgical site infections in patients who underwent abdominal surgery. Patients who will undergo abdominal surgery at Dr. Burhan Nalbantoğlu State Hospital will comprise the sample of volunteer patients who meet the inclusion criteria and agree to participate in the study. The data of the study was planned to be collected using the Patient Information Form, Surgical Site Infection Follow-up Form and Post Discharge Patient Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older
* Having undergone abdominal surgery
* Volunteering to participate in the research
* Patients without risk of preoperative malnutrition

Exclusion Criteria:

* Those who test positive for known Povidone Iodine allergy
* Those who use steroids and immunosuppressive drugs
* Those who used antibiotics due to infection in the last two weeks (prophylactic antibiotic use is not included in this item since all patients were given antibiotics for prophylaxis on the first day before surgery)
* Those diagnosed with Diabetes Mellitus (DM)
* Obese (BMI>30) patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection Follow-up Form | 30 days
  The primary outcome of this study was SSI within 30 days of surgery, as defined by the Centers for Disease Control and Prevention. Secondary outcomes were identification of the causative organism, and investigation of clinical factors such as body mass index (BMI), operation time, days of hospitalization, etc. that may be associated with SSI.

SECONDARY OUTCOMES:
Discharge Follow-up | 30 days
  All patients were followed up for SSI until discharge from hospital and at the outpatient visits. SSI surveillance data forms were used for the collection of primary and secondary outcome data.
  SSI rates and distribution of identified micro-organisms for each group will measured

CONTACTS AND LOCATIONS:
Overall Officials: Kerem Yıldız, PhD Student, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leaper DJ, Edmiston CE. World Health Organization: global guidelines for the prevention of surgical site infection. J Hosp Infect. 2017 Feb;95(2):135-136. doi: 10.1016/j.jhin.2016.12.016. Epub 2016 Dec 24. No abstract available. PMID 28139389
- [Background] Rogers SO Jr. Surgical Perspective: Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection 2017. Surg Infect (Larchmt). 2017 May/Jun;18(4):383-384. doi: 10.1089/sur.2017.097. No abstract available. PMID 28541803
- [Result] Gezer S, Yalvac HM, Gungor K, Yucesoy I. Povidone-iodine vs chlorhexidine alcohol for skin preparation in malignant and premalignant gynaecologic diseases: A randomized controlled study. Eur J Obstet Gynecol Reprod Biol. 2020 Jan;244:45-50. doi: 10.1016/j.ejogrb.2019.10.035. Epub 2019 Nov 9. PMID 31739120
- [Result] Wistrand C, Soderquist B, Nilsson U. Positive impact on heat loss and patient experience of preheated skin disinfection: a randomised controlled trial. J Clin Nurs. 2016 Nov;25(21-22):3144-3151. doi: 10.1111/jocn.13263. Epub 2016 Jun 3. PMID 27256458
- [Result] Wistrand C, Nilsson U. Effects and experiences of warm versus cold skin disinfection. Br J Nurs. 2011 Feb 10-23;20(3):148,150-1. doi: 10.12968/bjon.2011.20.3.148. PMID 21378634